CLINICAL TRIAL: NCT03927521
Title: Feasibility Study on the Use of PET-MRI / 68Ga-PSMA Imaging for HIFU-focal Treatment in the Event of Recurrent Prostate Cancer After Radiotherapy - PSMA Study
Acronym: PSMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0536
Record Dates: First submitted 2019-04-17; First posted 2019-04-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Post-Radiotherapy; Focal HIFU; PSMA; PET-MRI; Local recurrence
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focal HIFU guided by PET-MRI/68Ga-PSMA imaging (Experimental): Patient with local/focal prostate cancer recurrence after radiotherapy and no distant metastasis (negative PET-Choline imaging confirmed by PET-MRI/68Ga-PSMA) will be treated by Focal-HIFU
  Interventions: Procedure: Focal HIFU using PET-MRI/68Ga-PSMA imaging guidance

INTERVENTIONS:
Procedure: Focal HIFU using PET-MRI/68Ga-PSMA imaging guidance — Focal HIFU treatment will be conducted with the Focal One® device using the PET-MRI/68Ga-PSMA imaging. The treatment area will be defined using PET-MRI/68Ga-PSMA imaging data and 3D biopsies.

SUMMARY:
A significant proportion of patients with localized prostate cancer, and treated for curative intent by radiotherapy, have a local recurrence. Among these patients with local recurrence, few receive curative remedial treatment but most of them are treated with palliative hormonal therapy without any chance of long-term recovery.

The use of Focused Ultrasound (HIFU) in focal treatment (only on recurrence) is an effective and not very morbid option, especially compared to surgery. The quality of this treatment is conditioned by both an early diagnosis of recurrence, a precise localization of recurrence in the prostate and a rigorous extension assessment for the detection of occult metastases.

Innovations in medical imaging have led to the development of a new generation of "hybrid" machines that combine PET (Positron Emission Tomodensitometry) and MRI (Magnetic Resonance Imaging) technology. Associated with the use of 68Gallium-labeled PSMA (Prostate-Specific Membrane Antigen), a new tracer specific for prostate cancer, the investigators believe that this PET-MRI imaging technique can:

1. To identify at an early stage the metastatic patients and to allow a more adapted therapeutic management.
2. A better evaluation of the limits of local recurrence and therefore a more precise definition than with MRI alone of the tumor zone to be destroyed.

Finally, the investigators believe that the PET-MRI / 68Ga-PSMA exam, used for the selection of patients eligible for focal HIFU treatment and used for the treatment itself, should allow obtaining an optimal control of the cancer recurrence with the least possible side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years with a life expectancy of more than 5 years. Patients between the ages of 75 and 80 will need to have a G8 score > 14.
2. Biological recurrence after prostate radiotherapy confirmed with de Phoenix criteria (nadir + 2 ng/mL).
3. No prior or present evidence of lymph node metastasis, soft tissue metastasis or bone metastasis, assessed by the current radiographic exam (PET-Choline) AND the PET-MRI/68Ga-PSMA before Focal-HIFU.
4. Local prostate cancer recurrence confirmed by:

   * A multiparametric MRI showing a single tumor in the prostate gland at most 3 contiguous sextants confirmed by biopsies (Index tumor). Patients with multiple suspected MRI foci may be included if only one of these foci is confirmed by biopsies.
   * Index tumor confirmed by the PET-MRI/68Ga-PSMA.
5. PSA ≤ 10ng/ml.
6. Patient having been clearly informed of the study and having accepted, with sufficient reflection time, to participate by signing the informed consent form of the study.
7. Patient affiliated with health insurance or beneficiary of an equivalent plan.

Exclusion Criteria:

1. Contraindications to Focal-HIFU treatment.
2. Patient with a medical contraindication to Sonovue® injection.
3. Patient with a medical contraindication to MRI.
4. History of uncontrolled cancer and / or treated for less than 5 years (with the exception of basal cell skin cancer).
5. History of sclerosis of the bladder neck or urethral stenosis.
6. Patient at risk of bleeding according to medical advice. Patient with anticoagulants therapy must receive a treatment relay.
7. Patients with unstable neurological pathology.
8. Patient who has been treated for a therapeutic trial within 30 days of enrollment or who wishes to participate in an ongoing study that may interfere with this study.
9. Legal person protected by law.
10. Patient not able to understand the objectives of the study or refusing to comply with postoperative instructions.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Feasibility to use the PET-MRI/68Ga-PSMA imaging for Focal-HIFU guidance | At the time of the HIFU-focal treatment
  The feasibility to use the PET-MRI/68Ga-PSMA imaging for Focal-HIFU guidance will be evaluated by the possibility or not to use the target tumor contouring with the TEP-IRM au [68Ga]PSMA. This possibility will be determine for each patient with a systematic reviewing of TEP-IRM/[68Ga]PSMA and the target tumor contouring by 2 experts: a nuclear medicine specialist for TEP/[68Ga] PSMA and a radiologist, prostate MRI specialized.

SECONDARY OUTCOMES:
Interest of hybrid PET-MRI/[68Ga]PSMA imaging compared to PET-Choline for the metastasis detection during the initial assessment of first recurrence after radiotherapy. | Screening period.
  Interest of hybrid PET-MRI/[68Ga]PSMA imaging compared to PET-Choline for the metastasis detection during the initial assessment for first recurrence after radiotherapy will be evaluated by the proportion of patient who could not be treated by Focal-HIFU because of evidence of metastasis after the first PET-MRI/[68Ga]PSMA (screening failure rate).
Interest of hybrid PET-MRI/[68Ga]PSMA imaging compared to standard multiparametric MRI performed at the initial assessment AND 6 month after Focal-HIFU. | 6 months after focal HIFU therapy
  Interest of hybrid PET-MRI/[68Ga]PSMA imaging compared to standard multiparametric MRI will be evaluated by tumor volume comparison between both imaging method at the initial assessment AND 6 months after Focal-HIFU
Biological recurrence | 3 months and 6 months after focal HIFU therapy
  Biological recurrence will be evaluated by the proportion of biological recurrence, defined by a PSA nadir increase of more than 2 ng/mL at 3 and 6 months after Focal-HIFU.
Local control of tumor recurrence 6 months after Focal-HIFU guided by PET-MRI/[68Ga]PSMA imaging. | 6 months after focal HIFU therapy
  Local control of tumor recurrence 6 months after Focal-HIFU guided by PET-MRI/[68Ga]PSMA imaging will be evaluated by a second imaging assessment by PET-MRI/[68Ga]PSMA à 6 months after Focal-HIFU. In case of PSMA fixation on this imaging assessment, prostate biopsies will be performed.
Proportion of positives prostate biopsies | 3 months and 6 months after focal HIFU therapy
  Carcinologic evolution will be evaluated according to usual assessment performed for biological recurrence with proportion of positives prostate biopsies in the treated lobe and/or in the non-treated lobe.
Gleason score | 3 months and 6 months after focal HIFU therapy
  Carcinologic evolution will be evaluated according to usual assessment performed for biological recurrence with evolution of the Gleason score (4+3 = 7 or ≥ 8).
Extracapsular extension of prostate cancer. | 3 months and 6 months after focal HIFU therapy
  Carcinologic evolution will be evaluated according to usual assessment performed for biological recurrence with extracapsular extension of prostate cancer.
Metastatic free survival | Over the 6 months after focal HIFU therapy
  The metastatic free survival will be measured from the inclusion date to the date of first metastasis confirmation
QLQC30 score (Quality of life questionnaire) | 3 months and 6 months after focal HIFU therapy
  Quality of life will be assessed using the QLQC30 (Quality of Life questionnaire) questionnaire. It is a specific questionnaire to determine the quality of life a patient with cancer. It is composed of 30 questions with 4 potential answers going from: not at all, a little, enough or a lot, within 28 questions and with a visual scale going from 1 to 7 (7 being excellent and 1 being very bad) for the last 2 questions. The raw score is established by adding the score of each question and a linear transformation range it from 0 to 100. The higher the score, the better the quality of life.
EPIC-26 score (Urinary function questionnaire) | 3 months and 6 months after focal HIFU therapy
  Urinary function will be assessed using the EPIC-26 (The Expanded Prostate Cancer Index Composite) questionnaire. The EPIC-26 is a self-reported scale health-related quality of life questionnaire for prostate cancer patients. It is composed of 26 items in 4 different domains: urinary incontinence, urinary irritation/obstruction, bowel, sexual, and vitality/hormonal.
  Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale. Each items as a standardized value from 0 to 100. Then the average of the standardized value is determined in each domain to crate the summary score. The higher the score, the better the quality of life.
IPSS score (Urinary function questionnaire) | 3 months and 6 months after focal HIFU therapy
  Urinary function will be assessed using the IPSS (International Prostate Score Symptom) questionnaire. The IPSS questionnaire is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35. The score is then categorized as follow: Mild (symptoms score less than or equal to 7), Moderate (symptom score range 8-19), Severe (symptom score range 20-35). The higher the score, the worse the symptoms.
IIEF-5 score (Sexual function questionnaire) | 3 months and 6 months after focal HIFU therapy
  Sexual function will be assessed using will be assessed using the IIEF-5 (The International Index of Erectile Function) questionnaire.The IIEF-5 Questionnaire is composed of 5 items with 5 possible answers rating from 1 to 5 (very low, low, moderate, high, very high).
  The score is the sum of the ordinal responses to the 56 items. It is then categorized as follow: 22-25: No erectile dysfunction, 17-21: Mild erectile dysfunction, 12-16: Mild to moderate erectile dysfunction, 8-11: Moderate erectile dysfunction, 5-7: Severe erectile dysfunction. The higher the score, the better the sexual function.
Adverse event evaluation | During 6 months of follow-up after focal HIFU therapy
  Adverse events assessment between patient inclusion to the last study visit at 6 months (+/- 30 days) after Focal-HIFU treatment
Ancillary study: Measure of anti-tumoral immunity induction | Over the 6 months
  The consequences of HIFU treatment over immune anti-tumoral induction will be estimated by the description of Programmed death-ligand 1/ligand 2 (PDL1/L2) overexpression on immune cells and overexpression of Programmed cell death 1 (PD-1) on T lymphocytes (T-cells).
Circulating Tumor Cells (CTC) number | Over the 6 months
  The consequences of HIFU treatment over Messenger RNA (mRNA) will be estimated by measure of CTC number reduction (ancillary study).
ncRNA (non-coding RNA) PCA3 (Prostate cancer gene 3) level | Over the 6 months
  The consequences of HIFU treatment over PCA3 will be estimated by measure of ncRNA PCA3 level reduction (ancillary study).

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Urologie et Chirurgie de la Transplantation - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: RHU Perfuse web site — http://h5683.novius.net/